CLINICAL TRIAL: NCT01523704
Title: Comparison of the Safety and Efficacy of the Management of Pacemaker Patients Followed-up Via Home Monitoring vs. Conventional In-Office Follow-up
Brief Title: Safety and Efficacy Study of IPG Patient With Home Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik Japan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: atHome Study
Record Dates: First submitted 2012-01-26; First posted 2012-02-01 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Bradyarrhythmia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Monitoring(HM) (Experimental): Patients assigned to HM Group(HM follow-up ONLY) will have Home Monitoring programmed ON. They will be seen in the office for device interrogations at the 3-month follow-up, and at 27 month follow-up. In the meanwhile the device status will be evaluated using HM only for the 9, 15 and 21 month scheduled follow-up. Patients will visit the hospital for device interrogation on 27 month final follow-up.
  Interventions: Device: BIOTRONIK Home Monitoring System
- Control (Active Comparator): Patients assigned to Control Group (HM + Conventional In-office follow-up - Control group) will have HM programmed ON. In addition to HM, these patients will visit the hospital for device interrogation at 3, 9, 15, 21 and 27 month follow-ups.
  Interventions: Device: BIOTRONIK Home Monitoring System with In-office Follow-up

INTERVENTIONS:
Device: BIOTRONIK Home Monitoring System — Home Monitoring system transfers implantable device's data to the main server via internet.
  Arms: Home Monitoring(HM)
Device: BIOTRONIK Home Monitoring System with In-office Follow-up
  Arms: Control

SUMMARY:
The number of patients with implantable pulse generator (IPG) has steadily increased in Japan causing increment in number of in office follow-ups and greater burden on many hospitals.

The purpose of this multicenter randomized study is to demonstrate that BIOTRONIK Home Monitoring system reduces office follow-up visits without compromising patient safety.

DETAILED DESCRIPTION:
Patients will be randomized into HM follow-up only (Group 1) or HM & in-office follow-up (Group 2) and will be followed-up for 27 months.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for IPG implantation under Japanese guidelines
* Implanted within the last 45 days or being considered for implant with a BIOTRONIK IPG with Home Monitoring
* Able to utilize HM system throughout the study
* Ability to give informed consent
* Geographically stable and able to return for follow-ups for 27 months
* Over 20 years old
* Patient able to understand and follow the procedure stated in protocol

Exclusion Criteria:

* Contraindicated for IPG under Japanese guidelines
* Patients who are currently included in another cardiac clinical study
* Patients with expected life period of less than two years
* Patients who might undergo heart transplantation in next two years.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1327 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiichi Watanabe, MD, Principal Investigator — Fujita Health University
Locations (1):
- Fujita Health University, Toyoake, Aichi-ken, Japan

REFERENCES:
- [Derived] Watanabe E, Yamazaki F, Goto T, Asai T, Yamamoto T, Hirooka K, Sato T, Kasai A, Ueda M, Yamakawa T, Ueda Y, Yamamoto K, Tokunaga T, Sugai Y, Tanaka K, Hiramatsu S, Arakawa T, Schrader J, Varma N, Ando K. Remote Management of Pacemaker Patients With Biennial In-Clinic Evaluation: Continuous Home Monitoring in the Japanese At-Home Study: A Randomized Clinical Trial. Circ Arrhythm Electrophysiol. 2020 May;13(5):e007734. doi: 10.1161/CIRCEP.119.007734. Epub 2020 Apr 28. PMID 32342703

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1327 patients were enrolled. At the 3-month follow-up, 53 patients were excluded (24 withdrew consent, 17 death, 8 lost to follow-up and 4 protocol deviation). 1274 patients were randomized.
Groups:
- Home Monitoring Group: Patients assigned to HM Group(HM follow-up ONLY) will have Home Monitoring programmed ON. They will be seen in the office for device interrogations at the 3-month follow-up, and at 27 month follow-up. In the meanwhile the device status will be evaluated using HM only for the 9, 15 and 21 month scheduled follow-up. Patients will visit the hospital for device interrogation on 27 month final follow-up.
  BIOTRONIK Home Monitoring System: Home Monitoring system transfers implantable device's data to the main server via internet.
- Control: Patients assigned to Control Group (HM + Conventional In-office follow-up - Control group) will have HM programmed ON. In addition to HM, these patients will visit the hospital for device interrogation at 3, 9, 15, 21 and 27 month follow-ups.
  BIOTRONIK Home Monitoring System with In-office Follow-up
Period: Overall Study
Arm/Group | Home Monitoring Group | Control
Started | 636 (January 2012) | 638 (January 2012)
Completed | 558 (February 2016 (Enrollment: as of October 2013)) | 550 (February 2016 (Enrollment: as of October 2013))
Not Completed | 78 | 88

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Monitoring Group | Control | Total
Number analyzed (Participants) | 636 | 638 | 1274
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (9.7) | 77.2 (9.7) | 77 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297 | 345 | 642
  Male | 339 | 293 | 632
Region of Enrollment [Number; unit: participants]
  Japan | 636 | 638 | 1274

OUTCOME MEASURES:

1. Primary Outcome: Evaluation for Equivalence of the Number of Patients Who Meet the Composite Safety Endpoint Between Home Monitoring Group(HM) and Control Group Which is HM + Conventional In-office Follow-up
Description: The purpose of the primary endpoint is to compare the composite safety endpoint, Safety Event Rate (SER) which includes death, incidence of strokes and cardiovascular related serious adverse events requiring surgical interventions (e.g. device explants or lead revision) between HM Group and Control Group.
  Safety will be evaluated in the following testable hypothesis in an equivalence (non-inferiority) format:
  HØ: The safety event rate (SER) for a 24-month duration for Group 1 is not equivalent to the SER for Group 2.
  SER Group 1 - SER Group 2 ≥ Ha : The safety event rate (SER) for a 12-month duration for Group 1 is equivalent to the SER for Group 2 SER Group 1 - SER Group 2 < Where, ( )represents the allowable clinically significant difference. 5% was set for the study.
  A rejection of the null hypothesis (HØ) will indicate that the safety event rate for Group 1 is equivalent (non-inferior) to that of Group 2.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Home Monitoring Group | Control
Number analyzed (Participants) | 558 | 550
Participants | 61 | 65

2. Secondary Outcome: The Median (IQR) Numbers of In-office Follow-up（FU) Visits Per Patient-year
Description: Average numbers of outpatient follow-up(FU)s per patient are compared between Home Monitoring(HM) group and the control group, assessing total numbers of outpatient FUs combining regular and additional FUs. If the average number of visits in HM group is significantly less than that in Control group, it would serve as supporting evidence that the number of outpatient FUs can be reduced with HM.
  Analysis is performed on those patients that had a regular 3 months-FU following Intention to treat(ITT) principle. The analysis population of endpoint can be expected to be larger than the analysis population of the primary endpoints because patients with drop-out after the 3-months FU, but before the 27 months-FU will be included.
  The numbers of FU visits that occur in the 2 groups during the study period are compared as follows:
  AveN Group 1= Average number of FU visits per 2 years in the HM group AveN Control= Average number of FU visits per 2 years in the control group
Time Frame: 2 years
Population: 1134 patients were analysed, 534 from HM group and 600 from Control group. The lower number of patients from HM group can be explained by the fact that patients without any in-office FU after the 3M FU. Since HM group patients had no scheduled FUs after 3M before 27M, more patients of this group were excluded due to early drop-out.
Measure: Mean (Standard Deviation); unit: In-office FU visits per patient per year
Arm/Group | Home Monitoring(HM) | Control
Number analyzed (Participants) | 534 | 600
In-office FU visits per patient per year | 0.69 (0.43) | 2.00 (0.40)

3. Secondary Outcome: Efficacy of Home Monitoring：Average Cost for In-office Follow-up Per Patient-year
Description: The sum of insured medical expenses for regular and additional outpatient FUs will be compared between HM group and Control group. It shall include Fees of FU consultation, cardiac IPG instruction, and other diagnostic test , but treatment fees including medication. Hospitalization are not included.
  This analysis is performed on the same ITT population as the analysis set of the first secondary endpoint. To compensate for possible asymmetric drop-out, the comparison will not be cost per patient, but costs per patient-year.
  Study costs per patient will be calculated by summing up all relevant variables in 3mFU Randomization CRF (points2-11) as well as in InOffice FU CRF and in Additional InOffice FU CRF. Total costs per patient result by multiplying the sum of all points by 10. Unit measurement is Yen.
  H : The average costs in HM group are not less than that in Control group. AveCostsHM ≥ AveCostsControl Ha: The average costs in HM group are less than that in Control group.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Cost for in-office FU per patint-year
Arm/Group | Home Monitoring Group | Control
Number analyzed (Participants) | 635 | 634
Cost for in-office FU per patint-year | 21065 (23051) | 23552 (23986)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Home Monitoring Group | Control
All-Cause Mortality (participants affected / at risk) | 46/558 | 41/550
Serious Adverse Events (participants affected / at risk) | 68/558 | 68/550
Other Adverse Events (participants affected / at risk) | 7/558 | 16/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Monitoring Group (N=558) | Control (N=550)
The number of the composite primary endpoint (Cardiac disorders) | 61 (68) | 65 (68) — Composite primary endpoint: Death, Stroke and Cardiovascular surgery
The number of Stroke (Vascular disorders) | 8 (8) | 7 (7) — Details: Fatal and Non-fatal
The number of Cardiovascular surgery (Cardiac disorders) | 14 (14) | 20 (20) — Details: Coronary angioplasty, Ablation, Valve procedure, Other
Death (Cardiac disorders) | 46 (46) | 41 (41) — Details: Heart failure, Stroke, Other cardiovascular, Pulmonary, Cancer, Other non-cardiovascular, Unknown
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Monitoring Group (N=558) | Control (N=550)
Other safety events (Cardiac disorders) | 7 (7) | 16 (16) — Fracture/Fall and Syncope

LIMITATIONS AND CAVEATS:
We used one RM platform exclusively. This maintained continuous RM with 90.1% daily transmission success over two years, matching rates observed in other (shorter) trials. Whether our results are transferable to other RM platforms is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days